CLINICAL TRIAL: NCT01392066
Title: Psychosocial Adjustment of Patients and Their Partners Following Breast Cancer Diagnosis. A Prospective Cohort Study.
Brief Title: Psychosocial Adjustment of Patients and Their Partners Following Breast Cancer Diagnosis
Status: Completed | Type: Observational
Sponsor: University of Southern Denmark (Other)
Collaborators: Danish Cancer Society (Other); University of Groningen (Other); Rigshospitalet, Denmark (Other); Herlev Hospital (Other)
Responsible Party: Principal Investigator, Nina Rottmann, MSc, University of Southern Denmark
Other Study IDs: SDU-NFK-FK-2011; R40-A1920 (Other Grant/Funding Number: Danish Cancer Society); 2010-41-5193 (Other: Danish Data Protection Agency); 2012-41-0901 (Other: new ID from the Danish Data Protection Agency)
Record Dates: First submitted 2011-07-05; First posted 2011-07-12 (Estimated); Last update posted 2014-04-23 (Estimated); Status verified 2014-04

CONDITIONS: Breast Cancer
Keywords: breast neoplasms; spouses/partners; couples; interpersonal relations; psychosocial adjustment; psychological adaptation; depression; quality of life; dyadic coping; coping behavior; cohort; questionnaire
MeSH Terms: conditions — Breast Neoplasms; Depression | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Breast cancer patients and their partners: Patients with breast cancer and their cohabiting partners/spouses
  Interventions: Behavioral: questionnaire

INTERVENTIONS:
Behavioral: questionnaire — Both the patient and the partner/spouse fill out a questionnaire that assesses their psychosocial adjustment. Time for completion is ca. 30 minutes.
  The questionnaire is administered at baseline and 5- and 12-months follow up.

SUMMARY:
The purpose of this study is to describe psychosocial adjustment in patients with breast cancer and their cohabiting partners/spouses throughout the cancer trajectory, to study mutual influences of the partner on the patient and vice versa, and to identify risk and protective factors that influence the adjustment process in both patients and partners. The overall aim is to generate knowledge that helps enables us to integrate the partners' needs, problems and resources in treatment and rehabilitation of breast cancer patients.

DETAILED DESCRIPTION:
Breast cancer is a major life event. A patient's experience of breast cancer may depend heavily on her intimate partner. However, both patients and partners may experience depressed mood or other psychosocial adjustment problems. Individual and relationship factors, such as the couple's joint efforts to deal with the cancer experience, are likely to contribute to their psychosocial adjustment. More knowledge is needed on the adjustment problems patients and partners experience and how they deal with them.

The study investigates the following research questions:

* Which psychosocial adjustment problems do patients and partners experience throughout the cancer trajectory?
* To what extent do the patient's psychosocial adjustment problems influence the partner's psychosocial adjustment problems and vice versa?
* Which factors are associated with psychosocial adjustment problems?
* How do different strategies of dyadic coping influence the psychosocial adjustment of both the patient and the partner?

A prospective, population-based cohort will be established of women diagnosed with breast cancer in Denmark and their partners. The study combines questionnaire data and data from nationwide clinical and administrative registries.

An invitation letter and study material will be sent to patients by mail. Patients will be asked to invite their partner to participate in the study. Only couples in which both the patient and the partner wish to participate will be asked to complete the questionnaire at 5 and 12 months of follow-up.

Up to 3000 couples (3000 patients and 3000 partners) will be asked to participate in the study during the one year inclusion period.

ELIGIBILITY:
Inclusion Criteria:

* For patients: being a female patient diagnosed with primary breast cancer within the last four months
* For patients: cohabiting with a male partner/spouse
* For partners: being the male cohabiting partner/spouse of a patient diagnosed with primary breast cancer within the last four months

Exclusion Criteria:

* For patients: previous diagnosis of breast cancer or breast cancer relapse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: nationwide, population-based cohort of women diagnosed with breast cancer and their male cohabiting partner/spouse
Sampling Method: Probability Sample
Enrollment: 1584 (Actual)
Dates: Start 2011-07; Primary Completion 2013-07 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
quality of life | baseline
  self-report questionnaire SF-36
quality of life | 5-months follow up
  self-report questionnaire SF-36
quality of life | 12-months follow up
  self-report questionnaire SF-36
depressive symptoms | baseline
  self-report questionnaire CES-D
depressive symptoms | 5-months follow up
  self-report questionnaire CES-D
depressive symptoms | 12-months follow up
  self-report questionnaire CES-D
dyadic coping | baseline
  self-report questionnaire, Dyadic Coping Inventory and Ways of Providing Support Questionnaire
dyadic coping | 5-months follow up
  self-report questionnaire, Dyadic Coping Inventory and Ways of Providing Support Questionnaire
dyadic coping | 12-months follow up
  self-report questionnaire, Dyadic Coping Inventory and Ways of Providing Support Questionnaire

SECONDARY OUTCOMES:
illness perceptions | baseline
  self-report questionnaire Brief-Illness Perception Questionnaire
use of antidepressants | 12-months follow up
  registry information
work ability | baseline
  self-report item
work ability | 5-months follow up
  self-report item
work ability | 12-months follow up
  self-report item
sexual functioning | baseline
  self-report items (PROMIS item bank)
sexual functioning | 5-months follow up
  self-report items (PROMIS item bank)
sexual functioning | 12-months follow up
  self-report items (PROMIS item bank)
body image | baseline
  self-report questionnaire Body Image Scale
body image | 5-months follow up
  self-report questionnaire Body Image Scale
body image | 12-months follow up
  self-report questionnaire Body Image Scale
relationship functioning | baseline
  self-report items; quality of relationship and intimacy
relationship functioning | 5-months follow up
  self-report items; quality of relationship and intimacy
relationship functioning | 12-months follow up
  self-report items; quality of relationship and intimacy
symptom experience | baseline
  self-report questionnaire BCPT Eight Symptom Scale
symptom experience | 5-months follow up
  self-report questionnaire BCPT Eight Symptom Scale
symptom experience | 12-months follow up
  self-report questionnaire BCPT Eight Symptom Scale
partner's involvement in breast cancer | baseline
  self-report questionnaire
partner's involvement in breast cancer | 5-months follow up
  self-report questionnaire
partner's involvement in breast cancer | 12-months follow up
  self-report questionnaire
dimensions of sleep | 5-months follow up
  self-report questionnaire MOS sleep measure
dimensions of sleep | 12-months follow up
  self-report questionnaire MOS sleep measure

CONTACTS AND LOCATIONS:
Overall Officials: Dorte Gilså Hansen, MD, PhD, Study Chair — Research Unit of General Practice, Institute of Public Health, University of Southern Denmark; Christoffer Johansen, MD, PhD, DMSc, Study Chair — Institute of Cancer Epidemiology, Danish Cancer Society; Mariet Hagedoorn, MSc, PhD, Study Chair — University Medical Center Groningen; Nina Rottmann, MSc, Principal Investigator — Research Unit of General Practice, Institute of Public Health, University of Southern Denmark
Locations (1):
- University of Southern Denmark, Odense, Southern Denmark, Denmark